CLINICAL TRIAL: NCT06356909
Title: Study of PREMEdication Before Laryngoscopy in Neonates in France: a National Prospective Survey in French Neonatal Units and Neonatal Transport Teams
Brief Title: Study of PREMEdication Before Laryngoscopy in Neonates in France
Acronym: SUPREMEneo
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: SUPREMEneo
Record Dates: First submitted 2024-03-26; First posted 2024-04-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-04

CONDITIONS: Neonatal Respiratory Distress
Keywords: Sedo-analgesia; laryngoscopy; neonatal ICU; intubation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey of sedo-analgesia practices before laryngoscopy — The survey will evaluate adequation to the French best practice guidelines to improve their dissemination and to identify current practices of premedication before laryngoscopy in neonates in French units (agents, dosing, efficacy, safety)

SUMMARY:
This study is a national prospective survey on practices of premedication before laryngoscopy in neonates. The survey will evaluate adequation to the French best practice guidelines to improve their dissemination and to identify current practices of premedication before laryngoscopy in neonates in French units (agents, dosing, efficacy, safety)

DETAILED DESCRIPTION:
Laryngoscopy for intubation or less invasive surfactant administration (LISA) in neonates is a stressful and painful procedure that necessitates a sedo-analgesia except in the case of an immediate life-threatening emergency. Nevertheless, there are discrepancies in premedication practices amongst neonatal units. In order to optimize analgesia before laryngoscopy in neonates, the French neonatal society issued best practice guidelines in January 2023 for premedication before laryngoscopy in neonates. These guidelines were published in an English peer-reviewed journal and presented in national conferences. However, the implementation of new premedication protocols in neonatal units can be made difficult due to local habits, poor dissemination of the guidelines and a limited level of evidence on some premedication agents. Thus, conducting a survey one year after issuing the best practice guidelines on premedication seems important to evaluate French premedication practices and to evaluate the impact and dissemination of the guidelines

ELIGIBILITY:
Inclusion Criteria:

* Every neonate (corrected gestational age < 45 weeks of gestation) that undergoes a laryngoscopy (for intubation or LISA) or a laryngeal mask insertion, that received a premedication or not during the 28 days of the survey.

Exclusion Criteria:

* Laryngoscopy or laryngeal mask insertion in the operating room
* Opposition to data collection of a parent or holder of parental rights

Ages: 20 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Every neonate (corrected gestational age < 45 weeks of gestation) that undergoes a laryngoscopy (for intubation or LISA) or a laryngeal mask insertion, that received a premedication or not during the 28 days of the survey.
  The survey will be proposed to all French neonatal intensive care units (n=67), intensive care units (n=87) and pediatric transport teams (n=35) prior to the survey.
Sampling Method: Non-Probability Sample
Enrollment: 741 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who received a 1st sequence of sedo-analgesia consistent with best practice guidelines during laryngoscopy or laryngeal mask placement | Immediately after the laryngoscopy

SECONDARY OUTCOMES:
Molecules used for sedo-analgesia | Immediately after the laryngoscopy
Cumulative doses of sedo-analgesia used | Immediately after the laryngoscopy
Questionnaire for the operator describing reasons for non-compliance with best practice guidelines | Immediately after the laryngoscopy
Numeric rating scale for pain (by operator and assistant) | Immediately after the laryngoscopy
TRACHEA score (Tonus, Reactivity, Awareness & Conditions of intubation to Help in Endotracheal intubation Assessment) | Immediately after the laryngoscopy
  TRACHEA score from 0 to 10 where 0 represents adequate sedation with excellent conditions of intubation and 10 represents inadequate sedation with very poor conditions of intubation
Side effects related to the premedication | Immediately after the laryngoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Manon TAUZIN, MD, Principal Investigator — Centre hospitalier Intercommunal de Creteil
Locations (1):
- Centre Hospitalier Intercommunal de Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No